CLINICAL TRIAL: NCT04055753
Title: A Study to Assess Topoisomerase II Alpha (TOPO2A) as a Biomarker for Sensitivity to Doxorubicin/Doxil in Soft Tissue Sarcoma
Brief Title: Study to Assess TOPO2A as a Biomarker for Sensitivity to Doxorubicin/Doxil in Soft Tissue Sarcoma
Status: Active, not recruiting | Type: Observational
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: SAR-082
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — liposomal doxorubicin; Doxorubicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Doxorubicin
  Interventions: Drug: Doxorubicin
- Doxil
  Interventions: Drug: Doxil

INTERVENTIONS:
Drug: Doxil — Doxil 50 mg/m2, as per institutional standard
  Groups: Doxil
Drug: Doxorubicin — Doxorubicin 75 mg/m2, IV over 5-15 min OR Continuous infusion over 48-72 hours
  Groups: Doxorubicin

SUMMARY:
The primary aim of this study is to determine the utility of TOPO2A as a biomarker for sensitivity to doxorubicin or its derivatives. Patients whose planned therapy is doxorucibin or doxil single agent may be enrolled into this trial. In light of its recent FDA approval and differing mechanism of action, patients receiving olaratumab along with doxorubicin will be eligible for this study.

Doxorucibin will be administered at standard 21-day intervals. Doxil will be administered at standard 28-day intervals. Response to therapy will be assessed using standard RECIST criteria every 2 cycles. Patients will continue on study until disease progression, prohibitive toxicity or completion of cumulative dose of 450 mg/m2 of either agent. Overall survival will be assessed every 3 months for 1 year, every 6 months in year 2 and, annually until death.

ELIGIBILITY:
Inclusion Criteria:

* Patients must consent to providing tumor tissue prior to initiation of therapy if sufficient archival tissue is not available. Archival tissue is permitted if no other anticancer treatment was given after the tissue was obtained (not including surgery or radiation). If a biopsy is required, the treating physician should ensure that this can be done safely.
* Patients with STS will be eligible for the trial if their next planned chemotherapy will include single agent doxorubicin or doxil. Patients who will be receiving concomitant therapy with olaratumab will be allowed to participate.
* Sarcoma subtypes of angiosarcoma, epithelioid sarcoma, leiomyosarcoma, fibrosarcoma, myxofibrosarcoma, synovial sarcoma, pleomorphic rhabdomyosarcoma, undifferentiated pleomorphic sarcoma, liposarcoma (excluding well-differentiated) and malignant peripheral nerve sheath tumor will be included. These are subtypes for which a targeted therapy is not standard of care. All other subtypes will be included on a case by case basis as determined by the principle investigator.
* ≥ 18 years of age.
* Ability to understand and willingness to sign a written informed consent and HIPPA document
* Measurable disease by RECIST 1.1 criteria (at least one target lesion outside of previous radiation fields or progressed within a previous radiation field).
* Life expectancy of at least 3 months.
* All women of childbearing potential must have a negative serum pregnancy test and all subjects must agree to use effective means of contraception (surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 6 months after the last dose. Post-menopausal women must meet the criteria of 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >35 mIU/ml (IU/L).
* Patients must have normal organ and marrow function as defined below

  * Absolute neutrophil count > 1,500/mcL
  * Platelets > 100,000/mcL
  * Total bilirubin ≤ 1.5 X upper limit of normal (ULN)
  * AST/ALT (SGOT/SGPT) ≤ 3 X institutional normal limits; if liver metastases are present then ≤ 5 X ULN are allowed

Exclusion Criteria:

* Patients may not be receiving any other investigational agents, chemotherapy, radiation therapy or hormonal therapy (i.e. aromatase inhibitors for leiomyosarcoma), with the exception of olaratumab
* Pregnant or breast feeding women.
* Any concomitant medical issue that in the opinion of the treating physician would confound survival from sarcoma (e.g. other active cancer, symptomatic brain metastases, cardiac conditions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients whose planned therapy is doxorucibin or doxil single agent may be enrolled into this trial.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-08-12 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Best overall response | 6 years
  best response recorded from the start of the treatment until disease progression/recurrence

SECONDARY OUTCOMES:
Overall survival | 6 years
  defined as the time from initiation of treatment until death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States